CLINICAL TRIAL: NCT02285972
Title: Efficacy of Intravenous Dexketoprofen and Tenoxicam on Propofol Associated Injection Pain
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ordu University (Other)
Responsible Party: Principal Investigator, özgür yağan, MD, assistant professor, Ordu University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Odu-5
Record Dates: First submitted 2014-11-01; First posted 2014-11-07 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2014-11

CONDITIONS: Injection Pain
MeSH Terms: interventions — Sodium Chloride; dexketoprofen trometamol; tenoxicam

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor

ARMS (3):
- saline (Placebo Comparator)
  Interventions: Drug: saline
- dexketoprofen (Active Comparator)
  Interventions: Drug: dexketoprofen
- tenoxicam (Active Comparator)
  Interventions: Drug: tenoxicam

INTERVENTIONS:
Drug: saline — before the anesthesia induction, 2mL saline iv injection
  Other Names: serum physiologic
  Arms: saline
Drug: dexketoprofen — before the anesthesia induction, 50 mg (2mL) iv dexketoprofen
  Other Names: Arveles; Leodex
  Arms: dexketoprofen
Drug: tenoxicam — before the anesthesia induction, 20 mg (2mL) iv tenoxicam
  Other Names: Oksamen-L; Tilcotil
  Arms: tenoxicam

SUMMARY:
Propofol remains the most common drug for induction of general anaesthesia, although it causes considerable pain or discomfort on injection. Anesthesia providers have attempted a large number of remedies to prevent this pain on injection. Previously explored ideas include injecting propofol into larger veins, warming of the hand with hot packs, and intravenous pretreatment with numerous other medications. No studies to date have looked at the dexketoprofen and tenoxicam for the pretreatment of pain on injection caused by propofol. The investigators propose studying the use of dexketoprofen and tenoxicam for pretreatment of propofol related pain on injection.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists (ASA) physical status 1 and 2
* 18 - 65 years
* general anesthesia scheduled for elective surgery

Exclusion Criteria:

* age < 18 years, > 65 years
* pregnancy
* patients requiring a rapid sequence induction
* refusal to participate and patients already participating in another study
* allergy to study drugs
* communication difficulty
* psychiatric and neurolojic disorders
* use of analgesics or sedative drugs within 24 hours before surgery.
* emergency surgery
* history of drug or alcohol abuse
* ASA 3 and above

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2014-11; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Verbal Pain Score | Approximately one minute following administration of propofol.
Facial Pain Score | Approximately one minute following administration of propofol.

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology and Reanimation Dept. Ordu University Training and Research Hospital, Altinordu, Ordu, Turkey (Türkiye)